CLINICAL TRIAL: NCT03656913
Title: Validation of an Extremely Low Dose Computed Tomography Protocol for Diagnosing Urolithiasis in Children and Young Adults
Brief Title: Validation of Low Dose CT for Diagnosis of Urolithiasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-5183
Record Dates: First submitted 2018-08-31; First posted 2018-09-04 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Nephrolithiasis; Ureterolithiases
Keywords: Kidney Stone; Renal; Renal Stone
MeSH Terms: conditions — Nephrolithiasis; Ureterolithiasis; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Patients will receive both the clinically indicated and extremely low dose CT exams
  Interventions: Diagnostic Test: Extremely low dose CT

INTERVENTIONS:
Diagnostic Test: Extremely low dose CT — Patients undergoing clinically indicated CT will also receive the extremely low dose CT

SUMMARY:
The investigators have developed an extremely low dose renal computed tomography (CT) protocol that on preliminary testing has an effective dose in the range of a single view abdominal radiograph. The investigators plan to test this exam in patients with known or suspected urolithiasis undergoing clinically indicated CT.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and young adult patients (ages 4 to <21 years)
* Known or suspected urolithiasis
* Undergoing clinically indicated CT of the abdomen/pelvis

Exclusion Criteria:

* Pregnancy
* Prior enrollment in the same study (no patient will be enrolled more than once)

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of extremely low dose CT | Immediate
  Sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Trout, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center Burnet Campus, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No data sharing